CLINICAL TRIAL: NCT02783248
Title: French National Observatory of Percutaneous Mitral Commissurotomy (PMC) Immediate Score, Scanner, Late Results
Brief Title: French National Observatory of Percutaneous Mitral Commissurotomy
Acronym: CALCIMIT
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 15542
Record Dates: First submitted 2016-05-19; First posted 2016-05-26 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Mitral Stenosis
Keywords: Percutaneous mitral commissurotomy; Mitral Stenosis
MeSH Terms: conditions — Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mitral Stenosis: No specific protocol intervention occurs. All the cares are made as done usually.
  Patients who may be included are all consecutive patients who agreed to participate in the study and having a PMC in a French medical-surgical centers that perform more than 5 year PMC.
  All patients undergoing echocardiography with the realization of the score Wilkins and Cormier.
  Will then be included to validate the result of late score that patients who had a good immediate result of the PMC defined by: mitral valve area ≥ 1.5 cm² and IM ≤ 2/4. Patients with a poor immediate result of the PMC will not be monitored as part of the study but their data will be collected for the description of the population and analysis of immediate results.
  Patients in the study will receive an annual monitoring as recommended, independently of the study.

SUMMARY:
The aim of this study is to validate prospectively the predictive score of late results about a diverse population recruited in France and to evaluate the contribution in predicting the outcome of the PMC scanner to study the mitral calcium score and the location of the calcifications.

DETAILED DESCRIPTION:
This is a multicenter prospective observational study conducted in French medico-surgical sites.

The Percutaneous Mitral Commissurotomy (PMC) is the standard treatment for Mitral stenosis (MS) in patients with rheumatic favorable characteristics. In Western countries the MS reaches older patients with less favorable characteristics, including the presence of mitral calcifications. Calcifications are a factor of poor outcome of the PMC. The scanner appears as a useful examination for their study but is not carried out systematically. The prediction of late results of the PMC is particularly important in patients with non-ideal characteristics which form a particularly heterogeneous population. A score of late results of the PMC on the wider western series was recently released but has not to date received external validation. In this score, prediction results was multifactorial, with a consideration of paramount clinical factors, but also a prognostic significance of mitral calcifications.

The validation of predictive score of late results of the PMC, with the analysis of calcifications, would better select patients who may best benefit from PMC and those for which the surgical management is preferred.

The aim of this study is to validate an external sample predictive score of the event-free survival in patients who have had a good immediate result of the PMC.

This study, purely observational, does not create any special procedure outside the patient's usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* This will include all consecutive patients with rheumatic MS referred for PMC
* Patients who agreed to participate in the study, with signed consent

Exclusion Criteria:

* Contraindication to the PMC
* Contraindication to non injected scanner for centers performing a scanner
* Patient Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who agreed to participate in the study and having a PMC in a French medical-surgical centers that perform more than 5 PMC annually.
  The estimated number of patients is 500 over a period of 3 years. The inclusion of patients in the study is performed in the center of the referent investigating physician liability
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Event free survival at 3 years | 3 years
  Measurement of event-free survival after good result of the PMC, observed in our study. The composite endpoint event-free survival is defined as: cardiovascular survival without reoperation on the mitral valve and patient in NYHA I-II at last follow

CONTACTS AND LOCATIONS:
Locations (1):
- Bichat Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Iung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). [Guidelines on the management of valvular heart disease (version 2012). The Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)]. G Ital Cardiol (Rome). 2013 Mar;14(3):167-214. doi: 10.1714/1234.13659. No abstract available. Italian. PMID 23474606
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD; ACC/AHA Task Force Members. 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 10;129(23):e521-643. doi: 10.1161/CIR.0000000000000031. Epub 2014 Mar 3. No abstract available. PMID 24589853
- [Background] Wilkins GT, Weyman AE, Abascal VM, Block PC, Palacios IF. Percutaneous balloon dilatation of the mitral valve: an analysis of echocardiographic variables related to outcome and the mechanism of dilatation. Br Heart J. 1988 Oct;60(4):299-308. doi: 10.1136/hrt.60.4.299. PMID 3190958
- [Background] Abascal VM, Wilkins GT, Choong CY, Thomas JD, Palacios IF, Block PC, Weyman AE. Echocardiographic evaluation of mitral valve structure and function in patients followed for at least 6 months after percutaneous balloon mitral valvuloplasty. J Am Coll Cardiol. 1988 Sep;12(3):606-15. doi: 10.1016/s0735-1097(88)80045-7. PMID 3403819
- [Background] Palacios IF. Percutaneous mitral balloon valvuloplasty. Does it really last as long and do as well as surgery? Adv Cardiol. 2002;39:100-13. doi: 10.1159/000058916. No abstract available. PMID 12060906
- [Background] Iung B, Cormier B, Ducimetiere P, Porte JM, Nallet O, Michel PL, Acar J, Vahanian A. Immediate results of percutaneous mitral commissurotomy. A predictive model on a series of 1514 patients. Circulation. 1996 Nov 1;94(9):2124-30. doi: 10.1161/01.cir.94.9.2124. PMID 8901662
- [Background] Dreyfus J, Cimadevilla C, Nguyen V, Brochet E, Lepage L, Himbert D, Iung B, Vahanian A, Messika-Zeitoun D. Feasibility of percutaneous mitral commissurotomy in patients with commissural mitral valve calcification. Eur Heart J. 2014 Jun 21;35(24):1617-23. doi: 10.1093/eurheartj/eht561. Epub 2014 Jan 6. PMID 24394379
- [Background] Bouleti C, Iung B, Himbert D, Messika-Zeitoun D, Brochet E, Garbarz E, Cormier B, Vahanian A. Relationship between valve calcification and long-term results of percutaneous mitral commissurotomy for rheumatic mitral stenosis. Circ Cardiovasc Interv. 2014 Jun;7(3):381-9. doi: 10.1161/CIRCINTERVENTIONS.113.000858. Epub 2014 Apr 29. PMID 24782197
- [Background] Palacios IF, Block PC, Wilkins GT, Weyman AE. Follow-up of patients undergoing percutaneous mitral balloon valvotomy. Analysis of factors determining restenosis. Circulation. 1989 Mar;79(3):573-9. doi: 10.1161/01.cir.79.3.573. PMID 2917388
- [Background] Ben-Farhat M, Betbout F, Gamra H, Maatouk F, Ben-Hamda K, Abdellaoui M, Hammami S, Jarrar M, Addad F, Dridi Z. Predictors of long-term event-free survival and of freedom from restenosis after percutaneous balloon mitral commissurotomy. Am Heart J. 2001 Dec;142(6):1072-9. doi: 10.1067/mhj.2001.118470. PMID 11717614
- [Background] Bouleti C, Iung B, Laouenan C, Himbert D, Brochet E, Messika-Zeitoun D, Detaint D, Garbarz E, Cormier B, Michel PL, Mentre F, Vahanian A. Late results of percutaneous mitral commissurotomy up to 20 years: development and validation of a risk score predicting late functional results from a series of 912 patients. Circulation. 2012 May 1;125(17):2119-27. doi: 10.1161/CIRCULATIONAHA.111.055905. Epub 2012 Mar 28. PMID 22456478